CLINICAL TRIAL: NCT03276715
Title: A Cohort Study of Prognostic Factors in Lung Cancer Patients With Malignant Pleural Effusion (MPE).
Brief Title: Prognostic Factors on Malignant Pleural Effusion
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Mei Sze, Doctor, The University of Hong Kong
Other Study IDs: UW 16-307
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Pleural Effusion, Malignant; Lung Cancer
Keywords: malignant pleural effusion; lung cancer
MeSH Terms: conditions — Pleural Effusion, Malignant; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malignant pleural effusion can occur in up to half of the patients with metastatic disease. It can cause shortness of breath to patients and so far there is no protocol on its management.

The study is looking at patients with malignant pleural effusion and aims to identify its prognostic factors.

Pleural fluid and blood analysis will be performed as in the standard of care and results will be collected at the start of diagnosis. This will not affect subsequent management plan. Patients' disease course will be followed up and progress data will be collected. Data will then be analysed to identify relevant prognostic factors.

DETAILED DESCRIPTION:
Malignant pleural effusion (MPE) is common, and is estimated to affect up to a half of patients with malignancy, either at the time or during subsequent clinical course after the diagnosis of malignancy. Lung cancer is the most common cause of MPE, followed by breast cancer, lymphoma, unknown primary genitourinary and gastrointestinal carcinoma. Pleural involvement indicates dissemination of malignancy and suggests a poorer prognosis and the median survival rate ranges from 3 to 12 months, with lung cancer showing the shortest survival among Caucasian cohorts. Patients with MPE frequently suffer from effusion related symptoms requiring therapeutic drainage. Conventionally, the options of therapeutic drainage of MPE include needle aspiration, and intercostal drain insertion with or without chemical pleurodesis. Needle aspiration allows quick relief of effusion and symptoms, though the volume of pleural effusion being aspirated with each attempt of needle puncture is limited to 1-1.5 litres, and repeated puncture involves risks of complications. Intercostal drain insertion will allow gradual drainage of large pleural effusion over days, but the shortcomings being the long hospitalization of at least a week, and the presence of trapped lung would preclude chemical pleurodesis for definitive fluid control. Up to 40% of MPE patients still require repeated pleural drainage procedure, even after Talc chemical pleurodesis. The much longer hospitalization period is considered unfavourable for patients with limited lifespan in terms of weeks or a few months, who would spend more time with their family. In recent few years, indwelling pleural catheter (IPC) has provided a relatively novel option of palliative MPE drainage, on an ambulatory out-patient setting. IPC has been reported to be cost-effective, in particular for patients with survival of less than 14 weeks. With the limited time span, it is important to balance between the aim of symptomatic relief and maintaining patient's quality of life. Invasive procedures and prolonged hospitalisation can cause great distress to patients. Predicted survival of patients with MPE would be important in informing the most suitable method for relieving MPE. Previous studies have identified relevant factors on prediction of survival in patients with malignant pleural effusion but so far, there is no data for Chinese patients. The LENT scoring system (pleural fluid lactate dehydrogenase, Eastern Cooperative Oncology Group performance score, neutrophil -to-lymphocyte ratio and tumour type) is a new validated prognostic score in malignant pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* malignant pleural effusion (MPE) due to lung cancer

Exclusion Criteria:

* workup of MPE (pleural fluid results, blood test results, or treatment history) not available
* Patients unwilling to join study (for prospective recruitment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective retrieval of list of subjects diagnosed to have malignant pleural effusion (MPE). Subjects diagnosed to have MPE who are under the care of Department of Medicine in Queen Mary Hospital, Hong Kong, will be invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Further pleural intervention | 3 years
  Rate of fluid recurrence requiring invasive pleural interventions

SECONDARY OUTCOMES:
Survival | 3 years
  survival of lung cancer patient with malignant pleural effusion

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Chiang, MBBS(HK), Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clive AO, Kahan BC, Hooper CE, Bhatnagar R, Morley AJ, Zahan-Evans N, Bintcliffe OJ, Boshuizen RC, Fysh ET, Tobin CL, Medford AR, Harvey JE, van den Heuvel MM, Lee YC, Maskell NA. Predicting survival in malignant pleural effusion: development and validation of the LENT prognostic score. Thorax. 2014 Dec;69(12):1098-104. doi: 10.1136/thoraxjnl-2014-205285. Epub 2014 Aug 6. PMID 25100651
- [Background] Anevlavis S, Kouliatsis G, Sotiriou I, Koukourakis MI, Archontogeorgis K, Karpathiou G, Giatromanolaki A, Froudarakis ME. Prognostic factors in patients presenting with pleural effusion revealing malignancy. Respiration. 2014;87(4):311-6. doi: 10.1159/000356764. Epub 2014 Jan 22. PMID 24457947
- [Background] Bielsa S, Salud A, Martinez M, Esquerda A, Martin A, Rodriguez-Panadero F, Porcel JM. Prognostic significance of pleural fluid data in patients with malignant effusion. Eur J Intern Med. 2008 Jul;19(5):334-9. doi: 10.1016/j.ejim.2007.09.014. Epub 2007 Nov 8. PMID 18549935
- [Background] Thomas R, Francis R, Davies HE, Lee YC. Interventional therapies for malignant pleural effusions: the present and the future. Respirology. 2014 Aug;19(6):809-22. doi: 10.1111/resp.12328. Epub 2014 Jun 19. PMID 24947955
- [Background] Lui MM, Fitzgerald DB, Lee YC. Phenotyping malignant pleural effusions. Curr Opin Pulm Med. 2016 Jul;22(4):350-5. doi: 10.1097/MCP.0000000000000267. PMID 27055073
- [Background] Davies HE, Mishra EK, Kahan BC, Wrightson JM, Stanton AE, Guhan A, Davies CW, Grayez J, Harrison R, Prasad A, Crosthwaite N, Lee YC, Davies RJ, Miller RF, Rahman NM. Effect of an indwelling pleural catheter vs chest tube and talc pleurodesis for relieving dyspnea in patients with malignant pleural effusion: the TIME2 randomized controlled trial. JAMA. 2012 Jun 13;307(22):2383-9. doi: 10.1001/jama.2012.5535. PMID 22610520

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT03276715/Prot_SAP_000.pdf